CLINICAL TRIAL: NCT02212158
Title: Diabetes Intervention Program for Adolescents With Persistent High HA1c
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Heather MacKenzie, Ph.D., C. Psych. Candidate, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2014:206
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; adolescents; HA1c; psychological intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- motivational interviewing group (Experimental): Motivational Group Intervention:
  Group therapy sessions will include 8 teen sessions that cover the following topics: acceptance of diabetes, family issues, division of diabetes management, communication and facilitating motivation and skill development to improve diabetes care. Motivational interviewing and cognitive behavioral techniques will be the therapeutic modalities used in sessions. Parents will be involved in 3 therapy sessions that cover topics regarding family functioning, division of responsibility and parenting strategies.
  Interventions: Behavioral: motivational interviewing group

INTERVENTIONS:
Behavioral: motivational interviewing group — Group therapy sessions will include 8 teen sessions that cover the following topics: acceptance of diabetes, family issues, division of diabetes management, communication and facilitating motivation and skill development to improve diabetes care. Motivational interviewing and cognitive behavioral techniques will be the therapeutic modalities used in sessions. Parents will be involved in 3 therapy sessions that cover topics regarding family functioning, division of responsibility and parenting strategies.

SUMMARY:
The purpose of this project is to assess the feasibility and efficacy of a new group therapy program for adolescents with Type 1 diabetes and compromised metabolic control (high A1c). This intervention is aimed at addressing issues frequently found to be associated with poor control: knowledge deficits, parental supervision, parent-teen communication and psychosocial barriers. In order to test this new group therapy program, adolescents' HA1c and psychosocial functioning will be monitored pre- and post-intervention. It is hypothesized that individuals who participate in the group therapy program will show an improvement in their HA1c levels and quality of life, self-efficacy, supportive behaviors from family members, readiness to make improvements in their diabetes care and decrease symptoms of depression.

DETAILED DESCRIPTION:
Basic Design:

This study will pilot a group therapy intervention for adolescents seen in the diabetes clinic who have had elevated HA1c's for at least 3 months. This group will be offered in fall of 2014. Group therapy sessions will include 8 teen sessions that cover the following topics: acceptance of diabetes, family issues, division of diabetes management, communication and facilitating motivation and skill development to improve diabetes care. Motivational interviewing and cognitive behavioral techniques will be the therapeutic modalities used in sessions. Parents will be involved in 3 therapy sessions that cover topics regarding family functioning, division of responsibility and parenting strategies. Participants will complete questionnaires measuring self-efficacy, family support, quality of life, readiness to change and symptoms of depression. Questionnaires will be administered at an initial assessment prior to participation in the group, at completion of the 8 week program, at a follow-up visit 2 months following the completion of the group and 1 year post-intervention. Questionnaires will take approximately 45 minutes to complete. HA1c levels will be evaluated for participants every 3 months as per regular clinic care. This intervention program will be offered to teens upon an elevated HA1c result.

Primary Outcomes:

HA1c levels will be tested every three months as per regular clinic care. Basic demographic information will be obtained from participants during the initial assessment for the group (age, family size, and date of diagnosis of diabetes).

Secondary Outcomes:

Psychosocial functioning will be evaluated pre- and post-intervention by having participants and their parents fill out the following questionnaires: Self-efficacy for Diabetes Scale (SED); Diabetes Quality of Life for Youths; Diabetes Family Behavior Scale; Beck Depression Inventory for Youth (BDI-Y); Diabetes Management Questionnaire; Child Behavior Checklist (Parent form); Low Blood Sugar Survey, and Children's Hope Scale.

ELIGIBILITY:
Inclusion Criteria:

* The therapy group will be composed of teens that currently have a documented history of elevated HA1c's that have persisted for at least 3 months
* Potential candidates for the group will be recruited from all the physician's caseloads in the clinic.

Exclusion Criteria:

* Patients with Type II diabetes
* Those who are medically unstable due to other medical conditions
* Those who refuse to participate will not be included in the study

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-04 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline HA1c at 6 months post baseline | Baseline, 6-months post baseline
Change from baseline HA1c at 3 months post baseline | Baseline, 3-months post baseline
Change from Baseline HA1c at 9 months post baseline | Baseline, 9-months post baseline
Change in Baseline HA1c at 12 months post baseline | Baseline, 12-months post baseline

SECONDARY OUTCOMES:
Change from baseline in Self-efficacy for Diabetes scale (SED) at 8 weeks | baseline, 8 weeks
Change from baseline in Self-efficacy for Diabetes scale (SED) at 16 weeks | baseline, 16 weeks
Change from baseline in Self-efficacy for Diabetes scale (SED) at 60 weeks | baseline, 60 weeks
Change from baseline in Diabetes Family Behavior Scale at 8 weeks | baseline, 8 weeks
Change from baseline in Diabetes Family Behavior Scale at 16 weeks | baseline, 16 weeks
Change from baseline in Diabetes Family Behavior Scale at 60 weeks | baseline, 60 weeks
Change from baseline in Beck Depression Inventory for Youth (BDI-Y) at 8 weeks | baseline, 8 weeks
Change from baseline in Beck Depression Inventory for Youth (BDI-Y) at 16 weeks | baseline, 16 weeks
Change from baseline in Beck Depression Inventory for Youth (BDI-Y) at 60 weeks | baseline, 60 weeks
Change from baseline in Diabetes Quality of LIfe for Youth at 8 weeks | baseline, 8 weeks
Change from baseline in Diabetes Quality of LIfe for Youth at 16 weeks | baseline, 16 weeks
Change from baseline in Diabetes Quality of LIfe for Youth at 60 weeks | baseline, 60 weeks
Change from baseline in Diabetes Management Questionnaire at 8 weeks | baseline, 8 weeks
Change from baseline in Diabetes Management Questionnaire at 16 weeks | baseline, 16 weeks
Change from baseline in Diabetes Management Questionnaire at 60 weeks | baseline, 60 weeks
Change from baseline in Child Behavior Checklist (Parent form) at 8 weeks | baseline, 8 weeks
Change from baseline in Child Behavior Checklist (Parent form) at 16 weeks | baseline, 16 weeks
Change from baseline in Child Behavior Checklist (Parent form) at 60 weeks | baseline, 60 weeks
Change from baseline in Low Blood Sugar Survey at 8 weeks | baseline, 8 weeks
Change from baseline in Low Blood Sugar Survey at 16 weeks | baseline, 16 weeks
Change from baseline in Low Blood Sugar Survey at 60 weeks | baseline, 60 weeks
Change from baseline in Children's Hope Scale at 8 weeks | baseline, 8 weeks
Change from baseline in Children's Hope Scale at 16 weeks | baseline, 16 weeks
Change from baseline in Children's Hope Scale at 60 weeks | baseline, 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heather MacKenzie, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Diabetes Resource for Children and Adolescence, Winnipeg, Manitoba, Canada